CLINICAL TRIAL: NCT07059962
Title: Sensor-based Congestion Alert for Events in Peritoneal Dialysis (SCALE-PD)
Acronym: SCALE-PD
Status: Recruiting | Type: Observational
Sponsor: Bodyport Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-ScalePD-01
Record Dates: First submitted 2025-06-24; First posted 2025-07-11 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Kidney Disease; Peritoneal Dialysis (PD); End Stage Kidney Disease (ESRD)
Keywords: kidney disease; peritoneal dialysis; fluid overload; heart failure
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic; Edema; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- PD Patients: Patients with kidney disease on peritoneal dialysis.
  Interventions: Device: Bodyport Cardiac Scale

INTERVENTIONS:
Device: Bodyport Cardiac Scale — The Bodyport Cardiac Scale captures several physiological signals, which are used to derive multiple biomarkers that reflect a user's hemodynamic and fluid status.

SUMMARY:
To explore the use of the Bodyport Cardiac Scale in predicting worsening of events due to fluid overload in patients with kidney disease on peritoneal dialysis.

DETAILED DESCRIPTION:
The objective of this study is to explore the utility of hemodynamic biomarkers measured by the Bodyport Cardiac Scale in predicting worsening events attributable to fluid overload among those with kidney disease on peritoneal dialysis. The study will explore individual biomarkers, as well as composite biomarker indices, such as the Congestion Index and a novel PD Index.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years or older
2. Able to speak and read English, or able to speak and read Spanish and has a caregiver or family member who speaks English and can provide assistance
3. Able to stand on two bare feet unassisted
4. Receiving automated peritoneal dialysis for the treatment of ESKD
5. Followed on the Vantive Sharesource Remote Patient Management Platform

Exclusion Criteria:

1. Undergoing or plan to undergo hemodialysis in the next 12 months
2. Have a life expectancy of less than 12 months
3. Are pregnant or plan to become pregnant during the next 12 months
4. Weigh greater than 375 lbs
5. Planned kidney transplant within the next 12 months
6. Have an implanted neurostimulator system

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females 21 years of age or older, with end stage kidney disease undergoing peritoneal dialysis.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity Analysis | 1 year
  Sensitivity for predicting usable PDE > 0.40 and an alert rate of < 4.3 alerts per patient-year.

SECONDARY OUTCOMES:
Peritoneal Dialysis (PD) Events | 1 year
  Collection of approximately 40 usable PD Events for model development and validation. These events are defined as urgent, unscheduled clinic visits or emergency department visits or hospital admissions for worsening fluid overload and initiation or intensification of treatment for fluid overload or termination of treatment due to fluid related cause.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Desert Cities Dialysis, Victorville, California
  - Southeastern Clinical Research Institute, Augusta, Georgia
  - aQua Research Institute, LLC, Houston, Texas

IPD SHARING:
Plan to Share IPD: No